CLINICAL TRIAL: NCT06560073
Title: Safety & Results of Peroperative and Intraoperative Intravenous Tranexamic Acid in Diabetic Macular Tractional Retinal Detachment Surgeries
Brief Title: Intravenous Tranexamic Acid in Diabetic Macular TRD Surgeries
Acronym: TXA-DMTRD
Status: Completed | Type: Observational
Sponsor: Ahalia Foundation Eye Hospital (Other)
Responsible Party: Principal Investigator, Dr. Saurav Mahajan, Director Retina, Ahalia Foundation Eye Hospital
Other Study IDs: 202101; U1111-1311-5449 (Registry Identifier: WHO UTN)
Record Dates: First submitted 2024-08-15; First posted 2024-08-19 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Diabetic Retinopathy; Macular Traction Retinal Detachment
Keywords: tranexamic acid; diabetes mellitus; macular TRD
MeSH Terms: conditions — Diabetic Retinopathy; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to learn about safety and results of peroperative and intraoperative intravenous Tranexamic acid for diabetic macular tractional detachment eye surgeries . The main question it aims to answer is:

Adverse events and their frequency? immediate postoperative bleeding incidence? effective vitrectomy time?

DETAILED DESCRIPTION:
all Patients who agreed and gave informed consent forsurgery as well as to be included in study were included

Patients injected INTRAVENOUS TRANEXAMIC ACID 500 mg diluted to 10 ml with normal saline slowly in immediate preoperative period Accordingly, whenever bleeding was anticipated before removing active taut membranes or when bleeder was noted TXA 0.5 g was added upto maximum of 2 g. In Chronic kidney Disease patients dose was kept as maximum of 1.5 g

data analysis pack of microsoft excel will be used for statistical analysis. descriptive statistics will be applied. wherever mean of continuous variables is to be compared among subgroups, unpaired students t test will be used. To find any relationship among continuous variables , pearsons correlation or multiple regression will be used from data analysis pack of microsoft excel.

ELIGIBILITY:
Inclusion Criteria:

* Eyes of Diabetic patients having Macular Tractional Retinal detachment confirmed on Indirect Ophthalmoscope or B scan when associated with Vitreous hemorrhage or Optical Coherence Tomography

Exclusion Criteria:

* Pregnancy, lactation, Oral Contraceptive use, within 6 months thromboembolic disease ,Underlying cardiac arrhythmia where anticoagulation is indicated ,Seizures Severe liver disease,previous history of variceal bleeding ,Allergic history to Tranexamic acid

Ophthalmic exclusion criteria Previous vitreoretinal surgery Combination of tractional and rhegmatogenous retinal detachment Coexisting macular hole Macular dystrophies Arterial or venous occlusions Age related macular degeneration Extensive macular scarring Posterior segment inflammation

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: diabetic patients having Macular tractional retinal detachment who visited Retina department, Ahalia foundation eye hospital, palakkad, underwent surgery and gave informed written consent to be included in study
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Number of systemic adverse events | intraoperatively and postoperatively 24 hours
  Safety of intravenous tranexamic acid

SECONDARY OUTCOMES:
Number of systemic adverse events in patients having Chronic kidney disease | intraoperatively and postoperatively 24 hours
  Safety of intravenous tranexamic acid in Patients also having Chronic Kidney Disease
Surgical time for vitrectomy | intraoperatively
  Surgical time for vitrectomy that is less view blurring because of intraoperative bleed
Any relation between intraoperative use of Tranexamic acid and labetalol | intraoperatively
  labetalol dose needed
Number of vitrectomies converted intraoperatively to bimanual technique | intraoperatively
  Highly complex surgeries
Number of surgeries in which retinectomy required | intraoperatively
  Instances where it bleeds profusely and surgery could yet be completed successfully
Number of surgeries in which Perfluorocarbon liquid had to be used | intraoperatively
  PFCL acts as third hand- denotes complexity of surgery
Number of surgeries in which Internal Limiting Membrane peeling done | intraoperatively
  ilm peeling done after staining retina with Brilliant blue
Number of eyes having preretinal bleed at the end of surgery | immediate postoperatively
  to find efficacy of Tranexamic acid in decreasing immediate post operative bleed
Visual acuity change after surgery | 6 months postoperatively
  improvement in visual acuity

CONTACTS AND LOCATIONS:
Overall Officials: RAJKUMAR MAHESHWARI, MS, Study Director — Ahalia Foundation Eye Hospital; SAURAV MAHAJAN, MS, Principal Investigator — Ahalia Foundation Eye Hospital; AANCHAL MAINGI, DNB, Principal Investigator — AHALIA DIABETES HOSPITAL
Locations (1):
- Ahaliafoundation Eye Hospital, Palakkad, Kerala, India